CLINICAL TRIAL: NCT01889927
Title: INSPIRE-CF: A Randomised Controlled Trial Investigating the Clinical and Economic Benefits of an Alternative Model of Physiotherapy Care for Children With Cystic Fibrosis
Brief Title: INSPIRE-CF: an Alternative Physiotherapy Model for Children With Cystic Fibrosis
Acronym: INSPIRE-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11AR13
Record Dates: First submitted 2013-06-11; First posted 2013-07-01 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Cystic Fibrosis
Keywords: exercise; physiotherapy; lung function; quality of life
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Control (No Intervention): Control Group (Arm 1): Children randomised to the control group will receive 24-months of current model of specialist CF care.
- Group 2: Exercise Intervention (Active Comparator): Intervention group (Arm 2): Children randomised to the intervention group will receive 24-months of current model of specialist CF care PLUS a weekly structured, individually prescribed and personally supervised exercise intervention at a local fitness facility or at school.
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — The exercise intervention will include aerobic, anaerobic, strength, core conditioning and stretching components.
  Arms: Group 2: Exercise Intervention

SUMMARY:
The primary aim of the research is to evaluate whether an alternative model of cystic fibrosis (CF) physiotherapy care can produce statistically significant improvements in clinical and patient reported outcomes, and whether this alternative model is economically advantageous and/or sustainable.

Children randomised to the control group will receive 24-months of current model of CF care at Great Ormond Street Hospital (GOSH).

Children randomised to the intervention group will receive 24-months of current model of CF care at GOSH PLUS a weekly structured, individually prescribed and personally supervised exercise intervention at a local fitness facility or at school. The exercise prescription will include aerobic, anaerobic, strength, core conditioning and stretching components.

The main objectives of the study are:

1. Determine differences, if any, in lung function between the two groups;
2. Determine differences, if any, in exercise capacity between the two groups;
3. Evaluate cost of care of alternate model of care versus current model of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented diagnosis of Cystic Fibrosis;
* Male or female aged 6 years or older at baseline and <17years old at the end of the 2-year study;
* Currently under the primary care of the GOSH CF Unit;
* Able to perform Spirometry with a baseline FEV1 percentage predicted of 40% or higher, as measured on at least 3 occasions in the previous year, during times of clinical stability (i.e. not during an exacerbation, and not during or within 2 weeks of intravenous antibiotics);
* The participant's parent or legal guardian must be able to give informed consent; assent will be sought from all children.

Exclusion Criteria:

* Patients who have had lung transplantation;
* Patients listed for lung transplantation;
* Clinically significant disease or medical condition other than CF or CF-related conditions that in the opinion of the multi-disciplinary clinical team, would compromise the safety of the patient;
* Orthopaedic impairment that compromises exercise performance;
* Mental impairment leading to inability to cooperate;
* Unable to understand both verbal and/or written instructions English. Children will need to be able to understand exactly what the physiotherapists are instructing them do, for safe and effective exercise training sessions. Information sheets and questionnaires are only available in English;
* Participants, parents or legal guardians who are unwilling to sign consent to participate in the study.

The following criteria will not exclude a child from participating in the study, but based on the hospital's exercise laboratory's infection control protocol, may preclude the participant from Cardiopulmonary Exercise Testing.

* Patients with Methicillin-Resistant Staphylococcus Aureus;
* Patients with Burkholderia Cepacia.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | Baseline, 6, 12 and 24-month intervals.
  Spirometry data will also to be collected at outpatient clinics, annual reviews and during hospital admissions.

SECONDARY OUTCOMES:
Peak oxygen uptake (VO2Peak) | Baseline, 12 and 24-month intervals
  Gold standard exercise test to determine peak oxygen uptake during exercise
10m-Modified Shuttle Walk Test | Baseline, 6, 12 and 24 months
  Field test to assess functional exercise capacity. Distance covered and incremental level changes are evaluated over time.
Lung Clearance Index | Baseline, 12 and 24 months
  Multiple breath washout test to evaluate for changes in small airways
Height, weight, body mass index measurements | Baseline, 6, 12 and 24 months
  Height, weight and body mass index will be measured at regular intervals to evaluate for changes in growth parameters
Cystic Fibrosis Questionnaire | Baseline, 12 and 24 months
  Disease specific questionnaire to evaluate changes in quality of life in cystic fibrosis
Cost of care | Baseline, 12 and 24 months
  Evaluate differences in cost of care between the current model of CF care and the alternative model of care; and cost per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sean J Ledger, BSc MSc, Principal Investigator — Cystic Fibrosis Unit, Great Ormond Street Hospital for Children NHS Foundation Trust; Eleanor Main, BA MSc PhD, Principal Investigator — Institute of Child Health, University College London
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom